CLINICAL TRIAL: NCT00637234
Title: Oxcarbazepine as an Adjunct of Antipsychotic Therapy in Acute Schizophrenia
Acronym: OXC-SCZ
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Dr. F. Markus Leweke, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXC-SCZ CTRI476BDE06
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2008-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Oxcarbazepine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Oxcarbazepine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxcarbazepine — Oxcarbazepine (OXC), 300 mg tablets, up to 600 mg three times daily
  Other Names: Trileptal FCT 300MG.002; Film-coated tablet; Batch No.: X208 0802; Code: 3750031.002; Date of manufacture: September 2002; Date of evaluation: May 2004
  Arms: 1
Drug: Placebo — Placebo, 300 mg tablets, up to 600 mg three times daily
  Other Names: TRL PLA FCT.005; Film-coated tablet; Batch No.: X207 0802; Code: 3750411.005; Date of manufacture: September 2002; Date of evaluation: May 2004
  Arms: 2

SUMMARY:
Over recent years an approach with the adjunctive administration of various anticonvulsant drugs has been discussed and a limited number of open and controlled studies were performed for carbamazepine, valproic acid, and lamotrigine. While the latter shows promising effects in the long run it has some handling difficulties in the acute treatment of acute psychotic exacerbations. Valproic acid has shown inconsistent effects in schizophrenia with no significant effects in a recent controlled study. Although still controversially discussed, carbamazepine was found to offer beneficial effects in the treatment of schizophrenia. Nonetheless, data on these effects are limited by small sample sizes or poor design of most of the respective studies. Furthermore, the complex pharmacological interactions of new atypical neuroleptics with carbamazepine underline the necessity of alternative strategies in adjuvant treatment of schizophrenia as well as in combined treatment of bipolar disorders with mood stabilizers and neuroleptics.

Oxcarbazepine (OXC) is a new anticonvulsant drug that acts as a pro-drug for the 10-monohydroxy metabolite (MHD), an active metabolite also of carbamazepine that is suggested to be responsible for most of its therapeutic actions. Therefore, the pharmacological action of OXC is very well comparable to carbamazepine whilst there are fewer unwanted side effects of OXC regarding eg. skin rush, and effects on blood compounds or cardiotropic effects.

The effects of OXC on cytochrome CYP3A4 and CYP3A5 are moderate and UDPGT is only slightly affected by OXC, which leads to less interaction with other compounds on a pharmacokinetical level.

In psychiatry, the few studies published until now report positive effects of OXC in bipolar disorders. With regards to our own clinical observations, OXC has shown potential beneficial effects as an adjunct in the treatment of schizophrenia as well that require further evaluation in a controlled study design.

DETAILED DESCRIPTION:
This is an explorative controlled study with Oxcarbazepine (OXC) as an adjunct in the acute treatment of schizophrenia. The study will be performed in subjects between 18 and 50 years of age with an acute schizophrenic or schizophreniform disorder according to DSM-IV. The study will be performed according to Guidelines for Good Clinical Practice (GCP).

The primary hypothesis of this study is that adjunctive treatment with OXC yields at least comparable efficacy regarding antipsychotic actions with lower doses of neuroleptics and consequently substantially fewer adverse events.

A randomised controlled, double blind study is intended. During a 6 weeks treatment trial two groups of patients will be basically treated with olanzapine (starting with 5 mg after one week with an optional, BPRS-controlled step by step increase of about 2,5 mg each following week). Patients will receive a placebo controlled adjunctive therapy with OXC (1800 mg/day). After the initial lead-in of OXC within 7 days (allowing lorazepam as comedication), treatment with olanzapine will be started. Based on biometric calculations, a drop out adjusted sample size of 222 inpatients will be necessary

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia or schizophreniform psychosis according to DSM-IV
* BPRS score > 36 and BPRS psychosis cluster > 12
* Ability to provide written informed consent
* Participants are required an adequate contraception

Exclusion Criteria:

* Any severe neurological or somatic disorder
* Other psychiatric disorders including addictive disorders
* Positive urine drug screening for any compound except benzodiazepines
* No pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-07; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Amount of Olanzapine Co-medication | 5 weeks

SECONDARY OUTCOMES:
BPRS | 6 weeks
Extrapyramidal symptoms | 6 weeks
Weight gain | 6 weeks
Prolactin levels in plasma | 6 weeks
ECG QT-C time elongation | 6 weeks
Neurocognitive performance | 6 week

CONTACTS AND LOCATIONS:
Overall Officials: F. Markus Leweke, MD, Study Director — University of Cologne
Locations (2):
- Germany (2):
  - Isar-Amper-Klinikum gemeinnützige GmbH, Klinik Taufkirchen (Vils), Taufkirchen (Vils), Bavaria
  - University of Cologne, Dept. of Psychiatry and Psychotherapy, Cologne, North Rhine-Westphalia

REFERENCES:
- See also: Related Info — http://www.ecnp.net